CLINICAL TRIAL: NCT00555035
Title: A Double-Blind, Randomized, Placebo-Controlled, Single Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1349572 in Healthy Subjects
Brief Title: GSK1349572 First Time in Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ING111207
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: GSK1349572,; healthy volunteers
MeSH Terms: interventions — dolutegravir

INTERVENTIONS:
Drug: GSK1349572

SUMMARY:
To determine safety, tolerability and pharmacokinetics of GSK1349572

ELIGIBILITY:
Inclusion criteria:

* The subject is healthy.
* Healthy as judged by a responsible physician with no clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* The subject is ≥18 and ≤55 years of age.
* The subject is male or female.
* A female is eligible to enter and participate in this study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

  * Has had a hysterectomy or
  * Has had a bilateral oophorectomy (removal of the ovaries) or
  * Has had a bilateral tubal ligation or
  * Is post-menopausal (a demonstration of total cessation of menses for ≥ 1 year from the date of screening visit). A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal state. For this study FSH levels ≥ 40mIU/mL are consistent with menopause. If a subject is on estrogen replacement and menopausal status is questionable, estrogen replacement should be discontinued for 2 weeks and then the subject rescreened, as estrogen replacement can suppress FSH.
* A male is eligible to enter and participate in the study if he is surgically sterile OR if he either agrees to abstain from sexual intercourse with a female partner or agrees to use a condom/spermicide, in addition to having his female partner use another form of contraception, such as an intrauterine device (IUD), occlusive cap (diaphragm or cervical/vault cap) with spermicide, oral contraceptives, injectable progesterone, subdermal implants, female condom, contraceptive patch, or contraceptive vaginal ring, or has had a tubal ligation or hysterectomy. These criteria must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight ≥ 50 kg (110 lbs.) for men and ≥ 45 kg (99 lbs.) for women and body mass index (BMI) between 18.5-29.9 kg/m2 inclusive.
* A signed and dated written informed consent is obtained from the subject prior to screening.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.

Exclusion criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History/evidence of symptomatic or asymptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV-1 antibody result.
* Has a history of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men (1 drink (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits) within 6 months of the screening visit.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* Has a history of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit.
* The subject has a positive pre-study drug and/or alcohol screen.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* History or presence of allergy or intolerance to the study drug or its components or drugs of its class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort and iron supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, or serum creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* History of significant renal or hepatic diseases.
* History of Gilbert's syndrome.
* Exclusion Criteria for 24-Hour Screening Holter:

  * Any symptomatic arrhythmia (except isolated extra systoles).
  * Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (≥10 consecutive beats), complete heart block).
  * Non-sustained or sustained ventricular tachycardia (defined as ≥ 3 consecutive ventricular ectopic beats).
  * Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], WPW syndrome etc.).
  * Sinus Pauses > 3 seconds.
  * 300 or more supraventricular ectopic beats in 24 hours.
  * 250 or more ventricular ectopic beats in 24 hours.
* Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, AV block [2nd degree or higher], WPW syndrome).
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (≥3 consecutive ventricular ectopic beats)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Blood levels of drug over 72 hours. Laboratory test results over 72 hours Vital signs, ECG results over 72 hours | 72 hours.

SECONDARY OUTCOMES:
Dose proportionality over 72 hours | 72 hours.
GSK1349572 PK parameters: absorption lag time (tlag), and apparent clearance (CL/F) following single dose administration.
AUC(0-¥), AUC(0-t), Cmax, and C24 following single dose administration at different doses for the assessment of dose proportionality.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States